CLINICAL TRIAL: NCT01726244
Title: Effectiveness of an Self-care Program in the Prevention of Admissions of Patients With Hospitalizations Potentially Avoidable: Randomized Clinical Trial
Brief Title: Self-care Program in the Prevention of Admissions of Patients
Acronym: AUTOCUID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Naiara Parraza Diez, main researcher, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AC-01
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2012-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Heart Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Habitual Clinical Practice
- Intervention Group (Experimental): Multidisciplinary intervention consisting in controlling disease and stress associated to it, and modifying eating habits. A Nurse, nutritionist and a psychologist will be the responsible of these educational sessions. it will be three educational sessions. Patients with a BMI lower than 20 or bigger than 30 will be receive a closer follow up by nutritionist. In addition, patients with a score of 9 or more in the Patients Health Questionnaire-9 questionnaire will be also a closer follow up with the psychologist.
  Interventions: Behavioral: Multidisciplinary Intervention

INTERVENTIONS:
Behavioral: Multidisciplinary Intervention — Health education sessions consisting in controlling disease and stress asociated to it, and modifying eating habits
  Arms: Intervention Group

SUMMARY:
One of the most cost effective intervention is to avoid unnecessary hospitalizations in the national health system. These unnecessary admissions are increasing for several years, reaching rates of over 30% in patients with chronic obstructive pulmonary disease (COPD) or heart failure at two months of hospital discharge. There is scientific evidence suggesting that a multidisciplinary intervention consisting in controling disease and stress associated with disease, and modifying eating habits could reduce the number of hospitalizations due to disease decompensation.

The main objective of the study is to assess the rate of readmissions at year of multidisciplinary intervention in patients with COPD and / or heart failure.

We will select 144 patients who will be randomized to two groups (control and intervention group) and they will be followed for 12 months through 4 visits (1 month, 3 months, 6 months and 12 months of hospital discharge).

Patients assigned to the intervention group will be receive three educational sessions (one of them will be imparted by nursing, another by the nutritionist and the last one by the psychologist). In addition, patients with a BMI <20 and / or> 30 will receive a closer monitoring by the nutritionist).

Patients assigned to the control group will receive usual care in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* Heart failure: heart failure in clinically stable with ≥ II degree of NYHA . 1 or more emergency admissions for the same diagnosis in the prior year

Exclusion Criteria:

* Mental states that make difficult the self-care: Class 295, 296, 297, 298, 300, 301, 304 and 316 (schizophrenic disorders, episodic mood, delusional other nonorganic psychosis, anxiety, dissociative and somatoform, personality, alcohol and drug dependencies)
* Congenital respiratory diseases or presence of other obstructive pulmonary diseases
* Patients participating in other research studies.
* Other diseases that can affect patients' medium-term survival
* Moderate to severe cognitive impairment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Readmission rate | 12 months
  in the twelve months following the intervention, according to the electronic record of the hospital

SECONDARY OUTCOMES:
Number of admissions to emergency service or number of visits to general practitioner's office or number of visits to emergency service | 12 months
time until the first admission to the hospital | it wil be measured at 12 months
time until first visit to general practitioner's office | it will be measured at 12 months
time until the first visit to emergency service | it will be measured at 12 months
Health related quality of life through several questionnaires | At month, 3, 6 and 12 months after discharge
  COPD Assessment Test (CAT), self efficacy scale in COPD patients, SORT Form-36, Patient Health Questionnaire-9, Minnesota Living with Heart Failure Questionnaire (MLHFQ), Physical Activity Questionnaire (IPAQ), Barthel Index, European heart failure self-care behaviour scale.

OTHER OUTCOMES:
HbA1c | at month, 3, 6 and 12 months
  glycated hemoglobin
Type B natriuretic peptide (BNP), blood pressure | At month, 3, 6 and 12 months of discharge
APACHE III INDEX, Functional Category of New York Heart Association (NYHA) | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Araba Universitary Hospital (Txagorritxu), Vitoria-Gasteiz, Alava, Spain